CLINICAL TRIAL: NCT05921851
Title: Exploration of Early Warning System of Cardiac Arrest and Early Intervention
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K2993-K23C0266
Record Dates: First submitted 2023-06-18; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cardiac arrest: Cardiac arrest group: Patients who experience cardiac arrest during emergency diagnosis and treatment will use the time of cardiac arrest as the event time.
  Interventions: Other: no intervention
- control: The patient did not experience sudden cardiac arrest during the emergency diagnosis and treatment period, and was treated at the 24-hour time window in the emergency roomCollect data and use the end of the window as the event time.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The high incidence rate, high Case fatality rate rate and high rate of neurological impairment of cardiac arrest pose a serious threat to the health of the whole population, and also bring a huge economic burden. In recent years, the "American Heart Association AHA Cardiopulmonary resuscitation and Cardiovascular Emergency Guide" has always emphasized the importance of "life chain" for the survival of patients with cardiac arrest. The hospital's survival chain emphasizes early warning recognition and activation of emergency response systems, immediate high-quality CPR, rapid defibrillation, advanced life support, and post arrest care. However, there is an urgent need for improvement and enhancement in all aspects of the chain of life for cardiac arrest. Millimeter wave radar can transmit radar signals that penetrate non-metallic substances such as clothing, detect the micro motion signals caused by human respiration and heartbeat, and then process the signals. By calculating the frequency or phase shift information in the radar echo, patient activity information can be obtained, achieving contactless and real-time detection of patient activity in the room. And it can achieve tracking of targets in scenarios where multiple people exist, while monitoring the physical signs of each target in real-time [7]; Our team has developed Cardiopulmonary resuscitation Quality Monitoring Index (CQI) and Cardiopulmonary resuscitation Ventilation Mode (CPRV) in the early stage, which are very helpful to monitor and improve the quality of Cardiopulmonary resuscitation; In recent years, the application of bedside echocardiography (PoCUS) in emergency has been significantly expanded. Although transthoracic echocardiography (TTE) can provide valuable diagnostic information for patients with cardiac arrest, it has important limitations in dynamic compression of Cardiopulmonary resuscitation. TEE can overcome many limitations of TTE, and the combination of the two can achieve visualization of resuscitation, Many signs of Cardiopulmonary resuscitation that had not been found before have been found. On the other hand, international guidelines recommend that the compression site of Cardiopulmonary resuscitation should be in the lower half of the sternum. However, research shows that there are great changes in the shape of the chest and the organizational structure directly below the compression site in normal people. The left ventricle is located in the lower quarter of the sternum, lower than the lower third of the sternum. When Cardiopulmonary resuscitation is carried out according to the current guidelines, only a small part of the ventricle is subjected to external compression, and for spinal deformity, obesity There is no corresponding research and recommendation for pregnant women and other special groups, and the extensive development of chest CT Iterative reconstruction provides the possibility of individualized evaluation. In addition, the COVID-19 in China has not yet been completely controlled. For patients suspected or confirmed to be infected with novel coronavirus, it is still challenging to carry out Cardiopulmonary resuscitation that may produce aerosols when wearing protective equipment. In summary, establishing a clinical decision-making system for the survival chain under the new situation and optimizing the survival chain process in the guidelines is of great significance for improving the survival rate and prognosis of patients with cardiac arrest, and is of great value for improving national health levels and reducing the economic burden on the government.

ELIGIBILITY:
Inclusion Criteria:

* Enter the emergency room/ICU ward of Peking Union Medical College Hospital during 2019.1-2022.1 and 2022.12-2023.12 (emergency room)Diagnosing non flowing patients
* Age ≥ 18 years old, regardless of gender.
* No sudden cardiac arrest occurred upon admission.
* Laboratory tests are available within 24 hours before cardiac arrest occurs.
* Be able to understand the research protocol and willing to participate in this study, and provide written informed consent (applicable to Prospective cohort study).

Exclusion Criteria:

* Stay time is less than 24 hours.
* Trauma patients.
* Patients with sudden cardiac arrest outside the hospital.
* Refuse to participate and sign the informed consent form (applicable to the Prospective cohort study part

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enter the emergency room/ICU ward of Peking Union Medical College Hospital during 2019.1-2022.1 and 2022.12-2023.12 (emergency room)Diagnosing non flowing patients
  * Age ≥ 18 years old, regardless of gender.
  * No sudden cardiac arrest occurred upon admission.
  * Laboratory tests are available within 24 hours before cardiac arrest occurs.
  * Be able to understand the research protocol and willing to participate in this study, and provide written informed consent (applicable to Prospective cohort study).
Sampling Method: Non-Probability Sample
Enrollment: 12500 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of cardiac arrest | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No